CLINICAL TRIAL: NCT00272571
Title: The Effects of External Counter Pulsation Therapy (ECPT) on the Number and Function of Circulating Endothelial Progenitor Cells in Patients With Angina Pectoris
Brief Title: The Effects of External Counter Pulsation Therapy on Circulating Endothelial Progenitor Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-02-2701-JL-CTIL
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2006-01

CONDITIONS: Coronary Artery Disease
Keywords: ECPT, endothelial progenitor cells
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: External counter pulsation therapy

SUMMARY:
The objectives of the study are to test the hypothesis that external counter pulsation therapy (ECPT) provides clinical benefit by improving the number and function of endothelial progenitor cells (EPCs) in peripheral blood of patients with angina pectoris.

DETAILED DESCRIPTION:
ECPT is a non-invasive approach for increasing blood flow to the heart in patients with myocardial ischemia. ECPT produces beneficial effects in coronary artery disease (CAD) patients. However, the exact mechanisms of ECPT action are not defined yet. Evidence has now accumulated that bone marrow-derived cells with angiogenic capability, termed EPCs, circulate in the blood of adults. EPCs possess the ability to home to sites of ischemia and contribute to neoangiogenesis.

We prospectively study CAD patients [Canadian Cardiovascular Society (CCS) angina class II-IV], before and after ECPT , and compare them with age- and sex-matched controls. Peripheral blood CD34+ cells, EPCs (CD34/VEGFR2+ cells), EPC colony forming units (CFUs) and brachial artery endothelial function is assessed prior to and after ECPT. Percent improvement in endothelium-dependent brachial artery flow-mediated dilatation (%FMD) is assessed using high-resolution ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* CCS angina class II-IV

Exclusion Criteria:

* aortic regurgitation
* acute myocardial infarction <3 months
* systemic hypertension >180/110 mm
* atrial fibrillation
* deep vein thrombosis
* phlebitis and hemorrhagic diathesis
* pregnancy
* abdominal aortic aneurism
* metastatic tumor

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-08; Study Completion 2006-01

PRIMARY OUTCOMES:
The number of circulating endothelial progenitor cells in peripheral blood (before and one week after treatment)

SECONDARY OUTCOMES:
Brachial artery endothelial function (before and one week after treatment)
CCS angina class (before and one week after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leor, Prof., Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Neufeld cardiac research institute, Sheba medical center, Tel Litwinsky, Israel